CLINICAL TRIAL: NCT04651764
Title: Transanal Resection of Rectal Lesions With the ColubrisMX Endoluminal Surgical System (ELS System)
Brief Title: Transanal Resection of Rectal Lesions With the ColubrisMX ELS System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by ColubrisMX due to its identification of irregularities in the conduct of the trial (not related to clinical safety or effectiveness of the device)
Sponsor: ColubrisMX (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX-CSP-CS003
Record Dates: First submitted 2020-10-22; First posted 2020-12-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Rectal Adenoma; Rectal Polyp; Rectal Lesion
Keywords: Rectal Adenoma; Rectal Polyp; Rectal Lesion; Endoscopic Submucosal Dissection; Robotic Surgery; Endoluminal Surgery; Transanal Minimally Invasive Surgery; Transanal Surgery; Resection
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Robotically assisted transanal endoluminal resection of rectal lesion (Experimental)
  Interventions: Device: ColubrisMX Endoluminal Surgical (ELS) System

INTERVENTIONS:
Device: ColubrisMX Endoluminal Surgical (ELS) System — Robotically assisted transanal endoluminal resection of rectal lesion using the ColubrisMX Endoluminal Surgical (ELS) System

SUMMARY:
This study is a prospective, single-arm, multi-center, open-label, staged clinical study.

Overall Objective:

1. To evaluate the safety and effectiveness of the ELS System in subjects undergoing transanal endoluminal procedures in the rectum and distal colon (up to 17 cm from the anal verge).
2. To validate a program for training surgeons and their teams to successfully use the ELS System.

DETAILED DESCRIPTION:
Endoscopic Mucosal Resection (EMR) is the current standard treatment for non-malignant colorectal polyps in the United States. Large colorectal polyps are most often removed piecemeal when using EMR, as en-bloc resection becomes increasingly challenging with increasing lesion size. The major drawback of EMR is its low en-bloc resection rate. The piecemeal nature of the resection hinders margin assessment, which consequently results in low R0 resection rates and causes uncertainty regarding the appropriate treatment plan for the patient going forward. This outcome results in surveillance colonoscopies at shorter intervals to evaluate for recurrence, which in turn, increases patient anxiety and poses a burden on the healthcare system. Endoscopic Submucosal Dissection (ESD) enables en bloc resection and therefore improved histopathological assessment of margins and has been reported to have highly improved R0 resection rates when compared with EMR. ESD is a common treatment option for large colorectal lesions in Asia; however, the technical difficulty and steep learning curve, which are mainly attributed to the lack of traction and countertraction capability, have resulted in low adoption of ESD in the United States.

The ColubrisMX Endoluminal Surgical (ELS) System represents a marked advancement in the removal of non-malignant colorectal lesions. Robotic-assisted instrumentation with bimanual dexterity allows for application of traction and counter-traction and closure of the defect via suturing, and enables the technically challenging, single-handed ESD procedure to be conducted via a two-handed, robotic-assisted, transanal endoluminal surgical approach. The ELS System consists of two main components: the Patient Cart and the Surgeon Console. This system gains access by means of a flexible overtube (Colubriscope) that can be manually inserted up to 17 cm into the distal colon. The ELS System provides full visualization of the surgical site and the ability to manipulate up to two surgical instruments and a robotic-assisted third-party flexible endoscope (Olympus GIF-XP190), which is referred to as the "videoscope". The ELS Surgical Instruments are robotically assisted with full triangulation and articulation with up to 7 degrees of freedom to provide enhanced dexterity in narrow endoluminal anatomy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22-80 years
2. BMI ≤ 40 kg/m2
3. ASA score ≤ 3
4. Subject agrees to participate in the study by giving signed informed consent
5. Benign lesion that is located ≤ 17 cm from the anal verge, such as adenoma, submucosal nodule, or polyp
6. Lesion size is ≤ 7 cm, with size determined according to the American College of Gastroenterology (ACGE) and the American College of Colon and Rectal Surgeons (ACCRS) guidelines as the dimension of the lesion that is greatest in extent.

Exclusion Criteria:

Preoperative:

1. Anatomy unsuitable for endoscopic visualization or endoluminal surgery
2. Prior radiation treatment for colorectal cancer
3. Subject diagnosed with ≥ T1 colorectal cancer
4. Subject with distant metastases
5. Subject requiring Total Mesorectal Excision
6. Untreated active infection
7. Vulnerable population (e.g., prisoners, mentally disabled)
8. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic interventions
9. Breastfeeding or pregnant, or intend to become pregnant during the course of the study
10. Currently enrolled in or discontinued within the last 30 days from a clinical trial of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
11. In the opinion of the Investigator, the subject is unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.
12. Subjects with immunosuppression drugs (chemotherapy) due to an increased potential for infection and poor healing
13. Subjects with a high cardiac or pulmonary risk (these subjects require clearance from a cardiologist and pulmonologist)
14. Subjects on preoperative blood thinners, i.e., coumadin or heparin, that cannot be weaned prior to surgery
15. History of inflammatory bowel disease

Intraoperative:

1. Existing stricture or anatomical blockage in lower GI tract preventing Colubriscope from reaching desired position.
2. Inadequate bowel prep.
3. Complex anatomical findings not feasible for endoluminal or partial thickness approach.
4. Lesion demonstrates characteristics indicative of cancer, such as failure to lift upon submucosal injection, or any other features that raise the Investigator's suspicion of cancer.
5. Confirmation that lesion is located further than the intended use of the ELS System (past 17 cm from the anal verge).

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
En Bloc Resection Rate (percent) | Intraoperative
  The En Bloc Resection Rate (percent) is defined as the percentage of target lesions that are excised in a single specimen.
R0 Resection Rate (percent) | 30 days
  The R0 Resection Rate (percent) is defined as the percentage of target lesions that have lateral and deep margins that are free of neoplasia under microscopic visualization.
Complication-Free Rate (percent) | 30 days
  The Complication-Free Rate (percent) is defined as the percentage of subjects free from complications graded as Clavien-Dindo ≥ III intraoperatively or postoperatively through Day 30.

SECONDARY OUTCOMES:
Conversion-Free Rate (percent) | Intraoperative
  The Conversion-Free Rate (%) is defined as the percentage of intended procedures that do not require conversion to another platform (e.g., TAMIS or TEM) or surgical modality (i.e., laparoscopic or open surgery) to achieve successful completion.
Adverse Events (percent) | 30 days
  Data on adverse events will be collected during and after surgery. Each adverse event will be evaluated to determine the severity, relationship to the investigational device, action taken with respect to the investigational device, outcome, etc. Adverse events will be classified as mild, moderate, severe, or life-threatening.
Readmission Rate (percent) | 30 days
  The Readmission Rate (percent) is defined as the percentage of subjects with readmission that can be linked to the resection procedure requiring an interventional procedure up to 30 days after surgery.
Reoperation Rate (percent) | 30 days
  The Reoperation Rate (percent) is defined as the percentage of subjects requiring reoperation that can be linked to the resection procedure up to 30 days after surgery.
Estimated Blood Loss (mL) | Intraoperative
  Estimated Blood Loss (mL) is the amount of intraoperative blood loss (up to the point of needing transfusion). Estimated Blood Loss will be categorized as Significant, if transfusion is required, or Not Significant, if transfusion is not required.
Subjects Requiring Transfusion (percent) | 30 days
  Subjects Requiring Transfusion (percent) is defined as the percentage of subjects requiring transfusion prior to discharge.
Length of Stay (days) | 30 days
  The Length of Stay (days) is the amount of days that the subject stays in the hospital related to the resection procedure.
Mortality (percent) | 30 days
  Mortality (percent) is the percentage of subjects with a mortality from any cause up to 30 days, regardless of whether it was device/procedure-related or not.
Fecal Incontinence (percent) | 30 days
  Fecal Incontinence (percent) is the percentage of subjects with clinically significant disturbance to fecal continence from preoperative baseline to postoperative Day 30.
Rate of Rectal Stricture/Stenosis (percent) | 30 days
  A proctoscopic exam will be performed to assess rectal stricture/stenosis at 30 days post-procedure. Incidence of rectal stricture/stenosis detected at or before this follow-up visit will be recorded.
Local Recurrence Rate (percent) (subjects with cancer diagnosis only) | 5 years
  In subjects with lesions upstaged to histologically confirmed cancerous lesions post-resection with the ELS System, local recurrence will be monitored via five-year follow-up according to NCCN rectal cancer guidelines. The rate of local recurrence (%) in these subjects will be recorded.
Disease Free Survival (percent) (subjects with cancer diagnosis only) | 5 years
  In subjects with lesions upstaged to histologically confirmed cancerous lesions post-resection with the ELS System, disease free survival will be monitored via five-year follow-up according to NCCN rectal cancer guidelines. The rate of disease-free survival (%) in these subjects will be recorded.
Overall Survival (percent) (subjects with cancer diagnosis only) | 5 years
  In subjects with lesions upstaged to histologically confirmed cancerous lesions post-resection with the ELS System, overall survival will be monitored via five-year follow-up according to NCCN rectal cancer guidelines. The rate of overall survival (%) in these subjects will be recorded.
Vital Signs | 30 days
  Vital signs will be collected at preoperative baseline and post operative Days 7 and 30.
Clinical Laboratory Assessments | 1 day
  Clinical laboratory parameters will be collected at preoperative baseline and at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Wilson, MD, Principal Investigator — University of Texas; Erik Askenasy, MD, Principal Investigator — University of Texas; Sam Atallah, MD, Principal Investigator — University of Central Florida; Ovunc Bardakcioglu, MD, Principal Investigator — University of Nevada, Las Vegas
Locations (3):
- United States (3):
  - EndoSurgical Center of Florida, Orlando, Florida
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Memorial Hermann Southeast Hospital, Houston, Texas